CLINICAL TRIAL: NCT03436823
Title: Does Nurse Semi - Structured Interview Added to a Repeated Transcranial Magnetic Stimulation Improve Patients With Major Depressive Disorder? A Single Center Study, Randomized, Controlled and Single Blind
Brief Title: Does Nurse Semi Structured Interview Added to a rTMS Improve Patients With Major Depressive Disorder?
Acronym: DESTIMCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC14_9783_DESTIMCARE
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R.TMS + nurse semi-structured interview (Experimental): Repeated Transcranial Magnetic Stimulation sessions associated with nurse semi-structured interview
  Interventions: Other: nurse semi-structured interview
- R.TMS + Music & Relaxation (Sham Comparator): Repeated Transcranial Magnetic Stimulation sessions associated with music listening & relaxation with eyes closed
  Interventions: Other: Music & Relaxation with eyes closed

INTERVENTIONS:
Other: nurse semi-structured interview — The first session of rTMS is D1. From the first meeting to D14 semi -structured interviews are set up
  Arms: R.TMS + nurse semi-structured interview
Other: Music & Relaxation with eyes closed — The first session of rTMS is D1. From the first meeting to D14 music & relaxation with eyes closed sessions are set up
  Arms: R.TMS + Music & Relaxation

SUMMARY:
Repeated Transcranial Magnetic Stimulation - R.TMS - is currently part of the treatment for depressive illness. This non-invasive technique is designed to stimulate certain areas of the cerebral cortex involved in this pathology. FDA approved this treatment in routine for depressive illness. R.TMS still remains in assessment. Due to the heterogeneity of methods and the weakness of the cohorts therapeutic superiority can not concluded .

Stimulation parameters remain numerous even if a consensus is beginning to emerge. The therapeutic target is the left dorso - lateral prefrontal cortex. The lack of efficacy is probably due of the inaccuracy. The empirically location of the target does not take into account the inter-individual anatomical differences. The neuronavigation is becoming widespread in routine clinical practice.

The referent nurse stays with the patient all along the rTMS sessions. His role is to set up treatment, to ensure the safety and the well-being of the patient. An rTMS session is an average of 30 minutes and is a very special moment to create a specific therapeutic relationship.

No study was conducted to evaluate the therapeutic relationship. The assumption is made that rTMS with a semi - structured interview provides a qualitative and quantitative clinical response greater than a semi - structured rTMS without this nursing care. The investigators therefore propose to patients not receiving a semi-structured interview to listen to music with eyes closed.

DETAILED DESCRIPTION:
Repeated Transcranial Magnetic Stimulation - R.TMS - is currently part of the treatment for depressive illness. This non-invasive technique is designed to stimulate certain areas of the cerebral cortex involved in this pathology. The Food & Drug Administration - FDA - approved this treatment in routine for depressive illness. R.TMS still remains in assessment. Due to the heterogeneity of methods and the weakness of the cohorts therapeutic superiority can not concluded . Stimulation parameters remain numerous even if a consensus is beginning to emerge. The therapeutic target is the left dorso - lateral prefrontal cortex. The lack of efficacy is probably due of the inaccuracy. The empirically location of the target does not take into account the inter-individual anatomical differences. The neuronavigation is becoming widespread in routine clinical practice.

The referent nurse stays with the patient all along the rTMS sessions. His role is to set up treatment, to ensure the safety and the well-being of the patient. An rTMS session is an average of 30 minutes and is a very special moment to create a specific therapeutic relationship. To our knowledge, no study was conducted to evaluate the therapeutic relationship. The assumption is made that rTMS with a semi - structured interview provides a qualitative and quantitative clinical response greater than a semi - structured rTMS without this nursing care. The investigators, therefore propose to patients not receiving a semi-structured interview to listen to music with eyes closed.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteers aged 18 to 70,
* With the diagnosis of major depression, recurrent under the criteria of DSM.V,
* With an unmodified antidepressant treatment for 3 weeks,
* With a MADRS score greater than or equal to 21,
* With or without neuronavigated rTMS sessions,
* Informed and who have signed a consent.

Exclusion Criteria:

* Patients with psychotic symptoms,
* With alcohol dependence or other substances abuse,
* With the strength criteria defined by the V stage for Classification of Thase & Rush,
* Hospitalized without consent / or under legal protection for major.
* With a high risk of suicide - item 10 of the MADRS> 3 in the absence of hospitalization,
* With contraindications to the practice of MRI or rTMS due to previous seizures, neurological disorders and / or neurosurgical, metal prosthetic presence or foreign bodies pacemaker type intraocular ferromagnetic material,
* Aged over 70 years due to cortical alteration,
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
score of the Montgomery-Asberg Depression Rating Scale | day 44
  The ratings should be based on a clinical interview moving from broadly phrased questions about symptoms to more detailed ones which allow a precise rating of severity. The rater must decide whether the rating lies on the defined scale steps (0, 2, 4, 6) or between them (1, 3, 5). It is important to remember that it is only rare occasions that a depressed patient is encountered who cannot be rated on the items in the scale. If definite answers cannot be elicited from the patients, all relevant clues as well as information from other sources should be used as a basis for the rating in line with customary clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Drapier, MD, Principal Investigator — Centre Hospitalier Guillaume Régnier,
Locations (1):
- CHGR, Rennes, France